CLINICAL TRIAL: NCT06593080
Title: Validation of Treatment Decision Algorithms for Childhood Tuberculosis At District Health Care Levels in Mozambique and Zambia - the Decide-TB Cluster-randomized Pragmatic Trial
Brief Title: The DECIDE-TB Trial; Validation of Treatment Decision Algorithms for Childhood Tuberculosis
Acronym: DTB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chishala Chabala (Other)
Collaborators: University of Bordeaux (Other); Instituto Nacional de Saúde, Mozambique (Other Government); ADERA (Unknown); University of Stellenbosch (Other); Imperial College London (Other); Institut de Recherche pour le Développement (IRD) (Unknown); University of Sheffield (Other); Ludwig-Maximilians - University of Munich (Other); Ministry of Health, Zambia (Other Government); Ministry of Health, Mozambique (Other Government); Eduardo Mondlane University (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor-Investigator, Chishala Chabala, Principal Investigator, University of Zambia
Organization: University of Zambia (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: DECIDE-TB
Record Dates: First submitted 2024-08-01; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Tuberculosis; Child Health; HIV; Severe Acute Malnutrition
MeSH Terms: conditions — Tuberculosis; Severe Acute Malnutrition

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (No Intervention): The District Hospitals and Primary Health Centres in study districts will implement TB diagnosis for children as per the current Standard of Care (control) in both countries . In Mozambique, the SOC is based on local algorithms which include: TB symptoms screening (TB contact history), HIV testing, Xpert testing on induced sputum (and stool), and a tuberculin skin test. Urine Lipoarabinomannan (LAM) is indicated for Children Living with HIV (CLHIV). No CXR is performed.
  In Zambia, the SOC is based on the Union desk guide algorithm which includes: TB symptom screening (TB contact history), HIV testing and Xpert testing on respiratory or stool samples. Urine LAM is indicated for CLHIV,Severe Acute Malnutrition, sepsis, immune-suppression; chronic kidney diseases and cancer. CXRs are performed depending on the facilities. Other tests and imaging are advised in presumed extrapulmonary TB cases. A confirmed TB diagnosis is made based on a positive Xpert or LAM test.
- The comprehensive TDA based approach (Experimental): Children will benefit from the country SOC as described in the control arm, plus the study intervention
  Interventions: Other: The comprehensive TDA based approach

INTERVENTIONS:
Other: The comprehensive TDA based approach — The intervention consists of implementing a comprehensive TDA-based approach for TB diagnosis and treatment decision-making, including shorter treatment for non-severe TB in children identified as TB presumptive cases through a CDSS. It will also include the management of high-risk groups. In practice, all sick children will be assessed using the WHO-suggested TDAs A with CXR (DH) and B without CXR (PHC). CLHIV and those hospitalised with SAM at DH will have further assessment and treatment decisions based on the PAANTHER and TB-Speed SAM TDAs, respectively.
  Clinical and microbiological assessment data will be incorporated into a CDSS to help with the clinical decision to initiate TB treatment. The CDSS will incorporate specific features and test results for high-risk group children based on the PAANTHER TDA and the TB-Speed SAM TDA and will incorporate the results of the severity assessment to guide the choice of TB treatment duration once children are diagnosed with TB.
  Arms: The comprehensive TDA based approach

SUMMARY:
The Decide-TB project aims to generate evidence for the implementation of a comprehensive Treatment Decision Algorithms (TDA) based approach for TB in children living in high TB burden and resource-limited countries, at District Hospital (DH) and Primary Health Centre (PHC) levels, and to facilitate the integration of this evidence within practices and policies.

This programmatic pilot led by the National TB Programs (NTP) will test a TDA-based approach integrating TB screening, diagnosis, treatment decision-making, and disease severity assessment for shorter treatment eligibility, for use at a lower level of healthcare. This TDA-based approach will be evaluated in a hybrid effectiveness implementation study based on a pragmatic stepped wedge cluster-randomized trial. The Decide TB project will be implemented at the district level, targeting five districts in each country. Each cluster in a district will be made up of one district hospital and six primary health centers. The study will develop a Clinical Decision Support System (CDSS) to operationalize the use of TDAs, and strengthen District Health Information Systems (DHIS2) to collect individual data, which will contribute to monitoring and evaluation, clinical mentoring, and supervision by the country's NTPs.

DETAILED DESCRIPTION:
The Decide-TB trial is a pragmatic cluster-randomized study utilizing a stepped wedge design to provide scientific evidence on a comprehensive TDA-based approach for TB screening, diagnosis, and treatment in children under 15 years at low healthcare levels in Zambia and Mozambique.

The trial's primary objective is to evaluate the effectiveness, feasibility, implementation, acceptability, costs, cost-effectiveness, and adoption of a TDA-based approach for childhood TB screening, diagnosis, and treatment decision-making under programmatic conditions at District Hospitals (DH) and Primary Health Centres (PHC) levels in these countries.

There are five specific objectives corresponding to the trial's research components:

1. To assess the effectiveness of the comprehensive TDA-based approach in increasing TB case detection in children as compared to the Standard of Care (SOC), and in providing good quality TB diagnosis and treatment decision (diagnostic accuracy and reliability of treatment decision for TB and shorter treatment).
2. To describe the implementation and the feasibility of using the comprehensive TDA-based approach, including associated digital tools, and to identify contextual determinants influencing implementation and contribute to improved implementation/adaptations throughout intervention delivery.
3. To assess preferences, acceptability, and perceived feasibility of using the comprehensive TDA-based approach, including associated digital tools, among end-users, beneficiaries, and key stakeholders.
4. To assess the costs from the health system and the beneficiary (parents/caregivers of children) perspective, the cost-effectiveness of using the comprehensive TDA-based approach, including associated digital tools, and the budget impact of scaling up the intervention.
5. To assess the factors and stakeholders that support or constrain the adoption of the comprehensive TDA-based approach as health policy at district level.

The intervention will be implemented as a programmatic pilot, following the National TB Programs' decision in Mozambique and Zambia to adopt a TDA-based approach in line with World Health Organisation's (WHO) conditional recommendations. Additionally, both the standard of care and the intervention will be implemented in a non-randomized district to document diagnostic accuracy throughout the trial. The Decide-TB trial is a hybrid effectiveness-implementation trial (type 2), assessing both the clinical intervention's effectiveness and the feasibility and utility of the implementation strategy.

Diagnostic accuracy of both the standard of care and the intervention will be evaluated in an additional district, which will transition to the intervention phase alongside the last district selected per the stepped wedge design. Aggregated data will be retrospectively collected over 12 months from all participating districts and health facilities.

The Decide-TB trial endpoints include effectiveness, acceptability, implementation, health economics, and health policy. Effectiveness endpoints include the proportion of children who started TB treatment, the time it takes to make a treatment decision, and the consistency of TDA results with final treatment decisions, among other factors. Acceptability endpoints consider user preferences and local social value, whereas implementation endpoints evaluate the practicality, fidelity, contextual aspects, and sustainability of the TDA-based method. Health economics endpoints include cost assessments, cost-effectiveness, and budget impact of scaling up the TDA-based approach vs the standard of care, while health policy endpoints look at key stakeholders' roles, practices, and policy translation processes.

ELIGIBILITY:
Inclusion Criteria:

* For TB screening, all symptomatic children <16 years entering the selected health facilities (DH and PHC) at either outpatient (OPD) or inpatient (IPD) departments, including children from high-risk groups, as well as children identified as contact of TB cases.
* For access to TB diagnostic services and TDAs, children aged below 16 years identified with presumptive TB, i.e. those with ≥1 systematic screening criteria, among the following:

  * Cough with a duration of >2 weeks,
  * Fever with a duration of >2 weeks,
  * Documented weight loss,
  * History of TB contact with any duration of cough, OR identified by the site clinician irrespective of the above criteria, especially presumed extra-pulmonary TB cases.

Exclusion Criteria:

* Non presumptive TB cases
* Adult patients
* Patients not in the selected district or facilities

Max Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30240 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness endpoints: Children initiated on TB treatment | Throughout the study, an average of 24 months
  Proportion of children started on treatment for TB among sick children attending care at participant health facilities for any health complaints

SECONDARY OUTCOMES:
Effectiveness endpoints: Children treated for TB among those with presumptive TB | Throughout the study, an average of 24 months
  Proportion of children treated for TB among those with presumptive TB, including children with microbiologically confirmed TB.
Effectiveness endpoints: TB treatment proportion in high-risk pediatric groups | Throughout the study, an average of 24 months
  Proportion of children from high-risk groups treated for TB (age <2 years, CLHIV, children with SAM) i) among all children from high-risk groups attending care, ii) among children from high-risk groups with presumptive TB.
Effectiveness endpoints: Microbiologically confirmed TB cases | Throughout the study, an average of 24 months
  Proportion of children with TB that are microbiologically confirmed (i.e. smear or Xpert or LAM positive), ratio of <5 to 5-14 years among children with TB, ratio of pulmonary TB to extrapulmonary TB (EPTB).
Effectiveness endpoints: Time to TDA assessment completion | From the start of intervention to the end of the project, an average of 21 months
  Time from presumptive TB identification to final TB treatment decision and access to TB diagnostic assessment defined as the proportion of children with presumptive TB having completed assessment with the TDAs and CDSS, including in high-risk groups.
Effectiveness endpoints: Concordance of TDA results and TB treatment decisions | From the start of intervention to the end of the intervention, an average of 21 months
  Concordance of the TDA result and the final TB treatment decision using the proportion of children wrongly initiated or not initiated on TB treatment defined as: i) children not started on TB treatment despite positive score; ii) children initiated on TB treatment despite negative score. Reasons for both decisions will be collected.
Effectiveness endpoints: Missed and over-diagnosed TB cases | From the start of intervention to the end of the intervention, an average of 21 months
  Proportion of missed TB cases (false negative) and over-diagnosed TB cases (unlikely TB with a positive score, i.e. false positive).
Effectiveness endpoints: Concordance of TB severity evaluation and treatment regimen decision | From the start of intervention to the end of the intervention, an average of 21 months
  Concordance of the severity evaluation and decision for short TB treatment regimen using the proportion of i) children with 4-month TB treatment regimen used despite severe disease as assessed by the clinical/CXR evaluation; ii) children with 6-month TB treatment regimen despite non-severe disease as assessed by the clinical/CXR evaluation.
Effectiveness endpoints: False positive and negative TB severity assessments | From the start of intervention to the end of the intervention, an average of 21 months
  Proportion of false positive and false negative TB severity assessments at low level of health care: i) children with non-severe disease according to clinical criteria despite severe disease as evaluated by expert CXR read; ii) children with clinically assessed severe disease despite non-severe disease as evaluated by expert CXR read.
Effectiveness endpoints: Non-severe TB cases initiated on shorter treatment | From the start of intervention to the end of the intervention, an average of 21 months
  Proportion of children with presumptive TB and with non-severe TB disease initiated on shorter TB treatment.
Effectiveness endpoints: TB treatment outcomes stratified by severity and regimen duration. | From the start of intervention to the end of the intervention, an average of 21 months
  TB treatment outcomes as defined per WHO (treatment success, cured, treatment completion, loss to follow-up, death, treatment failure) overall and stratified by severity and regimen duration.
Effectiveness endpoints: Deaths averted | From the start of intervention to the end of the intervention, an average of 21 months
  Number of deaths averted assessed through modelling.
Effectiveness endpoints: Child TB among all diagnosed TB cases, including adults | Throughout the study, an average of 24 months
  Number of adults with TB, including microbiologically confirmed TB, and proportion of all TB diagnosed that is child TB.
Acceptability endpoints: Preferences | Throughout the study, an average of 24 months
  Proportion of healthcare providers' preferences in delivering childhood TB screening, diagnosis, and treatment decision-making, comparing the comprehensive TDA-based approach vs. the Standard of Care (SOC) approach, as assessed by TB diagnosis questionnaire, a self-administered questionnaire, completed every 3months in both arms, by all healthcare providers involved in child care.
Acceptability endpoints: Local social value (users) | Throughout the study, an average of 24 months
  Proportion of healthcare providers' preferences/ alignment with values and perceived potential to impact on lived experience) of the comprehensive TDA-based approach, including associated digital tools, to users (healthcare providers) as part of their work duties in childhood TB care, assessed by questionnaires.
Acceptability endpoints: Local social value (beneficiaries) | Throughout the study, an average of 24 months
  Proportion of beneficiaries' (children and their caregivers receiving a diagnosis of TB) local social value of the comprehensive TDA-based approach, including associated digital tools, as assessed by interviews and group discussions
Acceptability endpoints:Health systems and socioeconomic factors | Throughout the study, an average of 24 months
  Number of health systems and socioeconomic factors influencing preferences and local social value of the comprehensive TDA-based approach, including associated digital tools, for users and beneficiaries, as assessed by questionnaires, interviews and group discussions
Implementation endpoints: Feasibility | From the start of intervention to the end of the intervention, an average of 21 months
  Feasibility of implementing and delivering the comprehensive TDA-based approach, including associated digital tools: health systems, logistical, managerial, challenges faced during implementation, and solutions found as assessed by the TB diagnosis questionnaire.
Implementation endpoints: Fidelity | From the start of intervention to the end of the intervention, an average of 21 months
  Fidelity to intervention delivery and to implementation strategies: adherence to intervention procedures and implementation guide/manuals, adaptations, quality of implementation and intervention delivery.Assessed based on project process data (for example number and regularity of support supervision visits achieved compared to what was planned); fidelity of intervention delivery will based on the TB diagnosis questionnaire (number of health care worker reporting using TDAs to diagnose TB in children).
Implementation endpoints: Contextual factors | From the start of intervention to the end of the intervention, an average of 21 months
  Number of contextual factors influencing intervention delivery and implementation (at Individual, facility, health systems and community-level): barriers and facilitators as assessed by questionnaires, interviews and group discussions.
Implementation endpoints: Sustained intervention delivery | 6 months post intervention
  Number of facilities reporting using TDAs for childhood TB diagnosis 6 months post intervention period as assessed by sustainability questionaries.
Health economics endpoints: Cost analysis 1 | Throughout the study, an average of 24 months
  Total TB care costs from the health system perspective.
Health economics endpoints: Cost analysis 2 | Throughout the study, an average of 24 months
  Unit cost per TB care activity (e.g. clinical assessment, CXR).
Health economics endpoints: Cost analysis 3 | From the start of intervention to the end of the intervention, an average of 21 months
  Total TB care costs of overdiagnosis (false positive)
Health economics endpoints: Cost analysis 4 | Throughout the study, an average of 24 months
  Total costs incurred by parents/caregivers for receiving child TB care
Health economics endpoints: Cost effectiveness; Modelled health impact measure 1 | Throughout the study, an average of 24 months
  Number of children treated for TB.
Health economics endpoints: Cost effectiveness; Modelled health impact measure 2 | Throughout the study, an average of 24 months
  Number of adults treated for TB.
Health economics endpoints: Cost effectiveness; Modelled health impact measure 3 | Throughout the study, an average of 24 months
  Number of deaths.
Health economics endpoints: Cost effectiveness; Modelled health impact measure 4 | Throughout the study, an average of 24 months
  Measure of healthy life lost, either through premature death or living with disability due to illness; Disability-Adjusted Life Years (DALYs)
Health economics endpoints: Cost effectiveness- Incremental cost 1 | Throughout the study, an average of 24 months
  Incremental number of children treated for TB.
Health economics endpoints: Cost effectiveness- Incremental cost 2 | Throughout the study, an average of 24 months
  Incremental cost per Death averted.
Health economics endpoints: Cost effectiveness- Incremental cost 3 | Throughout the study, an average of 24 months
  Incremental cost per DALY averted.
Health economics endpoints: Budget impact 1 | Throughout the study; an average duration of 24 months and extending up to 5 years after its conclusion.
  Cost of scaling up the comprehensive TDA-based approach nationally.
Health economics endpoints: Budget impact 2 | Throughout the study; an average duration of 24 months and extending up to 5 years after its conclusion.
  Cumulative number of children and adults treated for TB, lives saved, and DALYs averted during a 5-year scale-up.
Health Policy endpoints: Roles, practices and processes | Throughout the study, an average of 24 months
  Roles, practices and processes among implementers and decision-makers of the comprehensive TDA-based approach, including associated digital tools, at district-level.
Health policy endpoints: Translation mechanism | At the end of the project, after 24 months since the start of the project
  Mechanism of translation of the research results and evidence on the comprehensive TDA-based approach, including associated digital tools, into public policies and practices: experience and perceptions of key stakeholders at regional, national and district-level.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Marcy, Principal Investigator — University of Bordeaux; Chishala Chabala, Principal Investigator — University of Zambia; Joanna Orne-Gliemann, Principal Investigator — University of Bordeaux; James Seddon, Principal Investigator — Imperial College London
Locations (29):
- Zambia (29):
  - Chawama Urban Health Centre, Chingola, Copperbelt
  - Chiwempala Urban Health Centre, Chingola, Copperbelt
  - Kabundi East Urban Health Clinic, Chingola, Copperbelt
  - Kasompe Urban Health Centre, Chingola, Copperbelt
  - Muchinshi Rural Health Centre, Chingola, Copperbelt
  - Nchanga 1 Urban Health Centre, Chingola, Copperbelt
  - Nchanga North Referal Hospital, Chingola, Copperbelt
  - Allessandras Urban Health Centre, Luanshya, Copperbelt
  - Chaisa Urban Health Centre, Luanshya, Copperbelt
  - Fisenge Urban Health Centre, Luanshya, Copperbelt
  - Kawama Urban Health Centre, Luanshya, Copperbelt
  - Malaika Urban Health Centre, Luanshya, Copperbelt
  - Mikomfwa Urban Health Centre, Luanshya, Copperbelt
  - Roan Antelope General Hospital, Luanshya, Copperbelt
  - Thomson District Hospital, Luanshya, Copperbelt
  - Chipepo Rural Health Centre, Chirundu, Southern Province
  - Hachipilika Rural Health Centre, Chirundu, Southern Province
  - Jamba Rural Health Centre, Chirundu, Southern Province
  - Kapululira Rural Health Centre, Chirundu, Southern Province
  - Lusitu Rural Health Centre, Chirundu, Southern Province
  - Mtendere Mission Referal hospital, Chirundu, Southern Province
  - Sikoongo Rural Health Centre, Chirundu, Southern Province
  - Habulile Rural Health Centre, Kalomo, Southern Province
  - Kalomo District Hospital, Kalomo, Southern Province
  - Kalomo Urban Health Centre, Kalomo, Southern Province
  - Mawaya Urban Health Centre, Kalomo, Southern Province
  - Namwianga Urban Health Centre, Kalomo, Southern Province
  - Nkandanzovu Rural Health Centre, Kalomo, Southern Province
  - Siachitema Rural Health Centre, Kalomo, Southern Province

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be available after de-identification. Access to the IPD dataset for each specific publication will be provided upon request to the coordinating investigators and with approval by the study sponsors and scientific oversight committee.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Access to data will be given after the publication of the main study results based on global data
Access Criteria: Data can be requested by Decide-TB consortium members and partners, as well as external research groups. Data can be utilised for secondary studies of the Decide-TB project, country-specific analyses, contributions to individual data meta-analyses, and analyses unrelated to the Decide-TB project's study topic. The request for data access must be submitted to the publication committee together with a concept paper detailing the analysis or study's aims, how the data will be utilised, the list of data or material requested, and how the original authors will be credited. Once the application is granted, data will be shared in accordance to a data and/or material sharing agreement that secures the terms of use.